CLINICAL TRIAL: NCT01859299
Title: Microbiome and Ocular Inflammatory Disease
Brief Title: Intestinal Bacteria and Ocular Inflammatory Disease
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130072; 13-EI-0072
Record Dates: First submitted 2013-05-17; First posted 2013-05-21 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-11-24

CONDITIONS: Uveitis
Keywords: Oral Tolerance; Uveitis; AMD; Natural History
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Affected: Participants with various types of uveitis
- Healthy controls: Participants without uveitis

SUMMARY:
Background:

- Uveitis is a general term describing a group of inflammatory diseases of the eye. The causes of uveitis are not fully understood. Researchers want to look at bacteria in the body that might be related to the inflammation. They will study the natural bacteria present in the gut and intestines of people with and without uveitis to understand their potential role in these diseases.

Objectives:

- To study the intestinal bacteria in people with and without uveitis or ocular inflammatory disease.

Eligibility:

* Individuals at least 18 years of age who have uveitis or ocular inflammatory disease.
* Individuals at least 18 years of age without uveitis or ocular inflammatory disease to serve as healthy controls.

Design:

* Participants may have more than one study visit (approximately 2-4) to assess possible changes in microbiome composition associated with treatment or disease activity.
* At each visit, participants will have a full eye examination, including vision and eye pressure tests. They will provide blood samples for testing. Participants will also be provided a stool collection kit to take home. The samples may be sent or brought back to the clinic.
* Treatment will not be provided as part of this study.

DETAILED DESCRIPTION:
Objective: What precipitates ocular inflammatory episodes remains unknown, but a possible potentiating factor is the microbiome. The microbiome has become increasingly studied with the advent of new techniques, but these have not been applied to uveitis. We wish to evaluate microbiome composition in patients with the ocular inflammatory diseases uveitis who may be on standard therapy or receiving orally-administered tolerizing antigen therapy.

Study Population: A total of 200 participants may be enrolled in this study. Of those participants, the goal is to enroll 50 healthy controls and 150 with various types of uveitis.

Design: This is an observational, prospective, single-center study. Participants will receive a complete ocular examination with clinical testing as determined clinically and will provide stool and blood samples using a standardized method. Participants may have multiple visits and may provide multiple samples in order to evaluate changes in microbiota composition with disease status or treatment.

Outcome Measures: Alterations in bacterial diversity, microbiota composition and changes in relative abundance of various taxa or species will be analyzed between healthy volunteers and participants and between various types of uveitis. In addition, comparisons will be made between these findings and the immunome and metabolome.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion Criteria for Uveitis Participants

1. Participant must be 18 years of age or older.
2. Participant must have a diagnosis of:

   Uveitis (or ocular inflammatory disorder)
3. Participant must be able to undergo slit lamp biomicroscopy.
4. Participant must understand and sign the protocol s informed consent document.

Inclusion Criteria for Healthy Volunteers

1. Participant must be 18 years of age or older.
2. Participant must be able to undergo slit lamp biomicroscopy.
3. Healthy controls will be age-and sex-matched individuals with no personal history of uveitis or other rheumatologic/autoimmune diseases (such as arthritis, inflammatory bowel disease, type 1 diabetes mellitus, psoriasis, Sjorgren s syndrome or multiple sclerosis) and no current use of corticosteroids, disease modifying antirheumatic drugs (DMARDs) including those with antibiotic properties (e.g., gold salts, sulfasalazine, hydroxychloroquine, minocycline) or any immunomodulatory drugs.
4. Participant must understand and sign the protocol s informed consent document.

EXCLUSION CRITERIA:

Exclusion Criteria for Uveitis Participants

1. Participants who are unable to provide informed consent.
2. Recent (<3 months prior) use of any antibiotic therapy
3. Current consumption of probiotics
4. Current extreme diet (parenteral nutrition, macrobiotic diet, etc.)
5. Known gastrointestinal (GI) tract neoplasm
6. Recent GI tract infection (gastroenteritis, colitis, diverticulitis, appendicitis) within the last month
7. Chronic unexplained diarrhea
8. Participant has or had a significant active infection (an infection requiring treatment as determined by the investigator) that required systemic antibiotic treatment within the past three months
9. Participant has any GI tract surgery leaving permanent residua (e.g., gastrectomy; bariatric surgery; colectomy)
10. Participant has inflammatory bowel disease (IBD)
11. Participant is pregnant or lactating.

Exclusion Criteria for Healthy Volunteers

1. Recent (<3 months prior) use of any antibiotic therapy
2. Current consumption of probiotics
3. Current extreme diet (parenteral nutrition, macrobiotic diet, etc.)
4. Known gastrointestinal (GI) tract neoplasm
5. Recent GI tract infection (gastroenteritis, colitis, diverticulitis, appendicitis) within the last month
6. Chronic unexplained diarrhea
7. Participant has or had a significant active infection (an infection requiring treatment as determined by the investigator) that required systemic antibiotic treatment within the past three months
8. Participant has any GI tract surgery leaving permanent residua (e.g., gastrectomy; bariatric surgery; colectomy)
9. Participant has inflammatory bowel disease (IBD)
10. Participant is pregnant or lactating.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 participants: 150 with uveitis; 50 healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2013-08-27 (Actual); Primary Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
The primary outcome is principal component analysis using the unweighted UniFrac distance metric of microbial composition; the significance between groups will be tested by the Adonis method (http://qiime.org/tutorials/category_comparison.html). | ongoing
  The primary outcome is principal component analysis using the unweighted UniFrac distance metric of microbial composition; the significance between groups will be tested by the Adonis method (http://qiime.org/tutorials/category_comparison.html).

SECONDARY OUTCOMES:
Abundance differences between groups at the level of individual phylotypes | ongoing
  Abundance differences between groups at the level of individual phylotypes (at different taxonomic levels, from phylum to species); the significance between groups will be tested using ANOVA
Abundance of microbial modules | ongoing
  abundance of microbial modules, constructed from microbial abundance co-occurrence networks and weighted gene co-expression network analysis (WGCNA) methodology, using the module eigenvector as the quantitative metric and statistically tested by ANOVA
Differences in lymphocyte and monocyte activation by different bacterial populations from the human microbiome results | ongoing
  Differences in lymphocyte and monocyte activation by different bacterial populations from the human microbiome results

CONTACTS AND LOCATIONS:
Overall Officials: Emily Y Chew, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nussenblatt RB, Gery I, Weiner HL, Ferris FL, Shiloach J, Remaley N, Perry C, Caspi RR, Hafler DA, Foster CS, Whitcup SM. Treatment of uveitis by oral administration of retinal antigens: results of a phase I/II randomized masked trial. Am J Ophthalmol. 1997 May;123(5):583-92. doi: 10.1016/s0002-9394(14)71070-0. PMID 9152063
- [Background] Presley LL, Ye J, Li X, Leblanc J, Zhang Z, Ruegger PM, Allard J, McGovern D, Ippoliti A, Roth B, Cui X, Jeske DR, Elashoff D, Goodglick L, Braun J, Borneman J. Host-microbe relationships in inflammatory bowel disease detected by bacterial and metaproteomic analysis of the mucosal-luminal interface. Inflamm Bowel Dis. 2012 Mar;18(3):409-17. doi: 10.1002/ibd.21793. Epub 2011 Jun 22. PMID 21698720
- [Background] Caporaso JG, Lauber CL, Walters WA, Berg-Lyons D, Lozupone CA, Turnbaugh PJ, Fierer N, Knight R. Global patterns of 16S rRNA diversity at a depth of millions of sequences per sample. Proc Natl Acad Sci U S A. 2011 Mar 15;108 Suppl 1(Suppl 1):4516-22. doi: 10.1073/pnas.1000080107. Epub 2010 Jun 3. PMID 20534432
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-EI-0072.html